CLINICAL TRIAL: NCT01118351
Title: Phase II Single Arm, Open Label, Single Institution Study of Continuous Sunitinib (Sutent) in Patients With High-Risk (BCG-Refractory) Superficial Transitional Cell Carcinoma (TCC) of the Bladder
Brief Title: Sunitinib Malate in Treating Patients With Recurrent Transitional Cell Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3808; NCI-2010-01137 (Other: NCI/CTRP); CASE 3808-CC530 (Other: Cancer Center IRB)
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Results first posted 2019-04-04 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Recurrent Bladder Cancer; Transitional Cell Carcinoma of the Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sunitinib; Immunohistochemistry; Microscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate; Other: immunohistochemistry staining method; Other: TdT-mediated dUTP nick end labeling assay; Other: light microscopy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sunitinib malate — Given orally
  Other Names: SU011248; SU11248; sunitinib; Sutent
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: TdT-mediated dUTP nick end labeling assay — Correlative studies
  Other Names: TUNEL assay
Other: light microscopy — Correlative studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib malate works in treating patients with recurrent transitional cell bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical efficacy of oral sunitinib (Sutent) given continuously for a maximum of 12 weeks, with respect to complete response rates at 12 months after completion of treatment in patients with high-risk superficial bladder cancer who have failed previous intravesical BCG.

SECONDARY OBJECTIVES:

I. To assess the impact of sunitinib treatment in recurrence-free survival, progression-free survival, and overall survival in patients with high-risk superficial TCC of the bladder who have failed previous intravesical BCG.

II. To evaluate the safety and tolerability of sunitinib (Sutent) administered in patients with high-risk superficial TCC of the bladder who have failed previous intravesical BCG.

TERTIARY OBJECTIVES:

I. To assess pre-treatment tissue baseline angiogenic markers and to evaluate the magnitude of the difference among these variables with post-treatment tumor tissue after treatment with sunitinib (Sutent).

II. To evaluate the effects of Sunitinib (Sutent) on immunosuppressive regulatory T cells (Tregs).

III. To determine the presence of circulating tumor cells in superficial BCG-refractory TCC patients.

OUTLINE:

Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion

* Patients must have clinically and histologically proven, recurrent superficial transitional cell carcinoma of the bladder after treatment with BCG therapy
* Patients could have received previous any INTRAVESICAL therapy including BCG and/or IFN and/or chemotherapy up to 3 years prior to registration
* Patients biopsy specimen should be available for review
* ECOG PS 0-1 (Karnofsky greater than 70%)
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8.5 g/dl
* Total bilirubin =< 1.5 X institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) =< 3.5 X institutional upper limit of normal
* Alkaline phosphatase =< 2.5 ULN ( =< 10 x ULN in presence of bone metastasis)
* Serum calcium of =< 12 mg/dl
* Creatinine =< 1.5 X institutional upper limit of normal
* INR =< 1.5, except for subjects receiving warfarin therapy
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of Sunitinib (Sutent) will be determined following review of their case by the Principal Investigator
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; sexually active patients must continue to use contraception for three months after completion of study therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* All patients must be informed of the investigational nature of this study and must provide written informed consent in accordance with institutional and federal guidelines

Exclusion

* Prior systemic chemotherapy for bladder cancer; all other systemic chemotherapy must have been completed at least 3 years prior to enrollment
* Prior treatment with any other anti-angiogenic therapy (including immunomodulatory agents such as thalidomide and lenalidomide, and anti-VEGF therapy with agents such as bevacizumab (Bevacizumab Avastin, Sunitinib (Sutent) and Sorafenib (Nexavar)
* Prior major surgery (not TURBT/Cystoscopy), radiation therapy, or systemic therapy within 4 weeks of starting the study treatment
* NCI CTCAE grade 3 hemorrhage within 4 weeks of starting study treatment
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
* Ongoing cardiac dysrhythmias of NCI CTCAE grade >= 2, or prolongation of the QTc interval to > 450 msec for males or > 470 msec for females (Atrial Fibrillation is allowed provided patients are rated controlled)
* Hypertension that cannot be controlled by medications
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) - related illness or infectious hepatitis type A, B or C
* Disease-free of prior malignancies for >= 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment
* Pregnancy or breastfeeding (Female patients must be surgically sterile or postmenopausal, or must agree to use effective contraception during the period of therapy; all female patients with reproductive potential must have a negative pregnancy test [serum or urine] prior to enrollment)
* Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy (The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-10; Primary Completion 2012-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Garcia, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - CCF-Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Derived] Zahoor H, Mir MC, Barata PC, Stephenson AJ, Campbell SC, Fergany A, Dreicer R, Garcia JA. Phase II trial of continuous treatment with sunitinib in patients with high-risk (BCG-refractory) non-muscle invasive bladder cancer. Invest New Drugs. 2019 Dec;37(6):1231-1238. doi: 10.1007/s10637-018-00716-w. Epub 2019 Jun 24. PMID 31231785

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I
Started | 19
Completed | 15
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: Years] | 72 [54 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Number of patients with complete response defined as negative cystoscopy with negative biopsy and no evidence of cancer on urine cytology 12 months after treatment with sunitinib.
Time Frame: At 12 months after completion of treatment
Population: All patients who received treatment and completed the 12 month follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 18
Participants | 4

2. Secondary Outcome: Recurrence-free Survival
Description: Time from registration (up to 28 days prior to treatment) to the first documentation of recurrence assessed up to 12 months after completion of treatment (up to 12 weeks). Time period can be up to 16 months from time of registration.
Time Frame: at 12 months after completion of treatment
Population: Patients that received treatment and completed follow up.
Measure: Median (Full Range); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 18
months | 3 [3 to 16]

3. Secondary Outcome: Progression-free Survival
Description: Number of patients last known to be alive and not to have progressed are censored at the last day of contact. Progression is defined as: Biopsy proven muscle invasive disease ≥ Stage T2 or death due to any cause.
Time Frame: at 12 months after completion of treatment
Population: All patients who received treatment and completed follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 18
Participants | 4

4. Secondary Outcome: Overall Survival
Description: Number of patients still alive from date of registration to date of death due to any cause.
Time Frame: at 12 months after completion of treatment
Population: All patients that received treatment and completed follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 18
Participants | 18

5. Secondary Outcome: Toxicity Assessed, Graded, and Tabulated Using CTCAE Version 3.0
Description: Number of participants that experienced adverse events.
Time Frame: at 12 months after completion of treatment
Population: All participants that received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 19
Participants | 19

6. Other Pre Specified Outcome: Immune Response
Description: The secondary outcome measure of response for the correlative studies will be the degree of apoptosis and the overexpression or not of known angiogenic markers (i.e. VEGF-R2, PDGF-R) an comparison by IHC analysis within bladder tumor tissue from the TURBT biopsy specimens with the post sunitinib (Sutent®) treatment TURBT specimens.
Time Frame: at 12 months after completion of treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Angiogenesis
Description: as for outcome 6
Time Frame: at 12 months after completion of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected while participants were on treatment (up to 12 weeks) and up to 1 year in follow-up.
Arm/Group | Arm I
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 3/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=19)
Cholecystitis (Hepatobiliary disorders) | 1
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 1
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 1
Hypertension (Cardiac disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils (Blood and lymphatic system disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=19)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (4)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (3)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (4)
Anorexia (Gastrointestinal disorders) | 7 (10)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 5 (9)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (6)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (3)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (7)
Cold Intolerance (General disorders) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 5 (5)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 13 (22)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Edema: head and neck (General disorders) | 1 (1)
Edema: limb (General disorders) | 5 (5)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 14 (22)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 5 (5)
Flu-like syndrome (General disorders) | 5 (7)
Cramps (Gastrointestinal disorders) | 1 (1)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 5 (8)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3 (3)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 12 (19)
Hemoglobin (Blood and lymphatic system disorders) | 12 (27)
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 2 (2)
Hemorrhage, GI - Varices (rectal) (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GU - Bladder (Renal and urinary disorders) | 1 (4)
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 1 (2)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypertension (Cardiac disorders) | 8 (10)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Bladder (urinary) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Mucosa (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1 (1)
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 2 (2)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 3 (3)
Insomnia (General disorders) | 4 (4)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 14 (22)
Lymphopenia (Blood and lymphatic system disorders) | 8 (20)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (2)
Mood alteration - Anxiety (Nervous system disorders) | 2 (2)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 3 (4)
Mucositis/stomatitis (functional/symptomatic) - Esophagus (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 8 (16)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Light/dark adaptation (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 8 (11)
Retinal tears (Eye disorders) | 1 (1)
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 (2)
Pain - Anus (Gastrointestinal disorders) | 1 (1)
Pain - Extremity-limb (General disorders) | 2 (3)
Pain - Head/headache (General disorders) | 1 (1)
Pain - Joint (General disorders) | 1 (1)
Pain - Middle ear (General disorders) | 1 (1)
Pain - Oral cavity (General disorders) | 1 (1)
Diffuse Arthralgia (General disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 17 (41)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (7)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 2 (3)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (6)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 7 (16)
Hemorrhage/Hematuria (Intermittent) (Renal and urinary disorders) | 1 (1)
Rigors/chills (General disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (7)
Stricture/stenosis (including anastomotic), GU - Urethra (Renal and urinary disorders) | 1 (1)
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1 (1)
Sweating (diaphoresis) (General disorders) | 1 (1)
Syndromes - Other (Cold) (General disorders) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 16 (21)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 2 (3)
Urine color change (Renal and urinary disorders) | 1 (1)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight loss (General disorders) | 2 (4)
Skin-Yellowing (Skin and subcutaneous tissue disorders) | 1 (1)
Tender Scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Greying/course hair (Skin and subcutaneous tissue disorders) | 1 (1)
Warm, tight "sunburn-like" skin (Skin and subcutaneous tissue disorders) | 1 (1)
GI (Other)-Dry Mucous Membranes, Nasal (Gastrointestinal disorders) | 1 (1)
Stomach "cramping" with flatulence (Gastrointestinal disorders) | 1 (1)
Visual disturbance (Eye disorders) | 1 (1)
Pain, Abdominal (Gas Cramps) (Gastrointestinal disorders) | 1 (1)
Pain, Chest (Gas Cramps) (Gastrointestinal disorders) | 1 (1)
Urinary, burning (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Accrual to the study was suspended and trial was prematurely closed due to a predefined futility rule that was part of the study's initial statistical design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes